CLINICAL TRIAL: NCT01227473
Title: A Mindfulness-based Intervention to Reduce Diabetes Risk in Pre-diabetic African Americans
Brief Title: We Can Prevent Diabetes: A Behavioral Intervention to Reduce Diabetes Risk in African Americans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Susan Gaylord, Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09-0563; 1R21AT004276-01A (Other: NIH NCCAM); 1R21AT004276-01 (NIH)
Record Dates: First submitted 2010-04-15; First posted 2010-10-25 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Prediabetes
Keywords: prediabetes; African Americans; mindfulness; behavioral; diabetes
MeSH Terms: conditions — Prediabetic State; Behavior; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mindfulness prediabetes education group (Experimental): The mindfulness-based diabetes prevention education group meets for 2 ½ hours per week for eight weeks, with one 4-hour retreat between the 6th and 7th weeks, and monthly booster sessions for 6 months. During the 8-week interventions, the group receives a 30-minute health behavior presentation (based on the landmark Diabetes Prevention Program). In the mindfulness-based diabetes prevention group, the instruction will be enhanced with instruction in mindfulness.
  Interventions: Behavioral: Mindfulness-based diabetes prevention education group
- conventional prediabetes education group (Active Comparator): The conventional diabetes prevention education group meets for 2 ½ hours per week for eight weeks, with one 4-hour retreat between the 6th and 7th weeks, and monthly booster sessions for 6 months. During the 8-week interventions, the group receives a 30-minute health behavior presentation (based on the landmark Diabetes Prevention Program). In the conventional diabetes prevention group, the instruction will be enhanced with group exercises and discussions.
  Interventions: Behavioral: Conventional diabetes prevention education group

INTERVENTIONS:
Behavioral: Mindfulness-based diabetes prevention education group — The mindfulness-based diabetes prevention group meets for 2 ½ hours per week for eight weeks, with one 4-hour retreat between the 6th and 7th weeks, and monthly booster sessions for 6 months. During the 8-week interventions, this group receives a 30-minute health behavior presentation (based on the landmark Diabetes Prevention Program). In the mindfulness-based diabetes prevention group, the instruction will be enhanced with a modified mindfulness meditation training designed to support the behavioral-change programming.
  Other Names: MBSR; DPP
  Arms: mindfulness prediabetes education group
Behavioral: Conventional diabetes prevention education group — The conventional diabetes prevention education group meets for 2 ½ hours per week for eight weeks, with one 4-hour retreat between the 6th and 7th weeks, and monthly booster sessions for 6 months. During the 8-week interventions, the group receives a 30-minute health behavior presentation (based on the landmark Diabetes Prevention Program). In the conventional diabetes prevention group, the instruction will be enhanced with group exercises and discussions.
  Other Names: DPP
  Arms: conventional prediabetes education group

SUMMARY:
Pre-diabetes, characterized by glucose levels that are above normal but below the diagnostic criteria for diabetes, is an increasingly common condition, particularly among African Americans. Changes in physical activity, changes in diet, and levels of stress influence the course of the disease. Helping individuals to reduce stress and to increase healthy coping strategies may enhance conventional diabetes prevention efforts, especially among African Americans. Mindfulness training is a cost-effective intervention which may be effective in reducing stress and enhancing the ability to make behavioral changes. This exploratory pilot study will examine the potential efficacy of a diabetes prevention education program that includes training in mindfulness-based stress reduction (intervention group) for pre-diabetic African Americans, comparing it to a conventional diabetes prevention program (control group) in the ability to improve glucose metabolism as well as other relevant physiological and psychological secondary outcomes.

DETAILED DESCRIPTION:
Pre-diabetes, characterized by glucose levels that are above normal but below the diagnostic criteria for diabetes, is an increasingly common condition affecting approximately 54 million U.S. adults. African Americans are disproportionately affected by pre-diabetes and experience high rates of diabetes-associated morbidity and mortality including damage to the circulatory system, kidneys, and nervous system. Patients with pre-diabetes who increase their physical activity and improve their diets have reduced risk of developing diabetes. Psychological distress negatively influences the course of the disease by increasing deleterious health behaviors; preventing scheduling and maintenance of positive behavior change; and stimulating HPA-axis activation and dysregulation, which may have a direct impact on insulin resistance and glucose metabolism. African Americans may have increased exposure to stress and increased vulnerability to adverse stress-related health outcomes like diabetes, because of their unique history, sociocultural experiences, and societal position in the U.S. Helping individuals to reduce stress and to increase healthy coping strategies may enhance conventional diabetes prevention efforts, especially among African Americans.

Mindfulness-based stress reduction (MBSR), a mind-body practice with a wide range of health benefits, has been shown to result in statistically significant reductions in psychological stress and anxiety in randomized, controlled studies. Mindfulness training is cost-effective in comparison with other small-group or individualized programs, and can be taught safely and effectively by well-trained instructors. There is little research, and no randomized, controlled trials of MBSR as a treatment for individuals with pre-diabetes. There is also little research on the acceptability of MBSR program to a prediabetic subgroup of African Americans, or on the acceptability of an MBSR program for a general population of African Americans.

Overall goals of this exploratory pilot study are to study the potential efficacy of a diabetes prevention education program that includes training in mindfulness-based stress reduction for pre-diabetic African Americans. Specific Aims are 1) to determine the feasibility of developing a clinical trial to compare the effectiveness of a mindfulness-based diabetes prevention program (treatment group) with a conventional diabetes prevention program (control group) in improving glucose metabolism in pre-diabetic African American adults; 2) to identify relevant physiological and psychological secondary outcomes associated with a mindfulness-based, educational self-care program in African-Americans with pre-diabetes; 3) to assess the acceptability and cultural relevance of MBSR for pre-diabetic African Americans via a post-intervention qualitative study, to include interviews of participants, dropouts, and instructors; and 4) to identify, and find solutions for, problems in conducting a well-powered clinical trial to assess the efficacy of a mindfulness-based diabetes prevention program in improving glucose metabolism in pre-diabetic African-Americans.

ELIGIBILITY:
Inclusion Criteria:

* African-American
* 25-65 years of age
* meeting the ADA criteria for pre-diabetes (either by fasting plasma glucose (FPG) of 100-125 mg/dl or glucose of 140-199 mg/dl at 2 hours in an oral glucose tolerance test (OGTT))or a HbA1c of 5.7-6.4%
* experiencing some degree of stress
* willing to attend 1 1/2 hour group meetings once weekly for 8 weeks, followed by monthly booster sessions for six months, and to complete assessment instruments.

Exclusion Criteria:

* diabetes diagnosed by a physician
* past or current use of hypoglycemic medication (except gestational diabetes)
* disease associated with disordered glucose metabolism
* use of medications associated with impaired glucose metabolism
* active treatment for or history of a major medical illness
* previous training in meditation or mindful yoga, tai chi, qigong
* pregnant or planning a pregnancy

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
insulin resistance, as measured by the homeostatic model assessment-insulin resistance (HOMA-IR) | Fasting samples will be collected 3 weeks, on average, before the intervention and at 3 months post intervention.
  The homeostatic model assessment-insulin resistance (HOMA-IR) is a calculated measure based on the FPG and fasting insulin levels.

SECONDARY OUTCOMES:
Salivary cortisol | Salivary cortisol will be measured before the intervention and at 2 weeks, 3 months, and 6 months post intervention
Insulin resistance as measured by the HOMA-IR | 2 weeks and 6 months post-intervention
  The HOMA-IR is calculated from the fasting insulin and fasting glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Gaylord, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States